CLINICAL TRIAL: NCT02648022
Title: Integrated Care for Patients With High Risk Substance Use and Psychiatric Disorders With Chronic Hepatitis C Receiving Direct Acting Antiviral Treatment
Brief Title: Integrated Care for Patients With High Risk Substance Use and Psychiatric Disorder With Chronic Direct Acting Antiviral Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: IIR 07-101-A
Record Dates: First submitted 2015-12-21; First posted 2016-01-06 (Estimated); Results first posted 2016-05-20 (Estimated); Last update posted 2016-05-20 (Estimated); Status verified 2016-05

CONDITIONS: Hepatitis C; Depression; PTSD; Substance Use Disorder; Fibrosis
Keywords: Care Integration; Hepatitis C; Substance Use Disorder; PTSD
MeSH Terms: conditions — Hepatitis C; Depression; Stress Disorders, Post-Traumatic; Substance-Related Disorders; Fibrosis | interventions — Case Management

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Integrated Care (Experimental): Consisted of brief mental health interventions and case management provided in a collaborative treatment environment.
  Interventions: Behavioral: Brief mental health interventions and case management
- Usual Care (No Intervention): The usual care group received "standard of care" required for HCV patients as currently performed in each clinic. All usual care patients were evaluated by their HCV Clinic treatment team, usually consisting of clinical nursing staff, the treating physician, and a clinic psychiatrist or psychologist

INTERVENTIONS:
Behavioral: Brief mental health interventions and case management — The mental health practitioner (MHP) provided brief interventions and follow up sessions designed to reduce the risk factors that are barriers to successful antiviral treatment (substance use, depression, PTSD. Second, MHP provided ongoing case management services to these patients, with an emphasis on navigating the complex HCV care process, preparation for antiviral treatment, and managing the treatment process (adherence, side effects, etc). Third, the MHP also activated the patient and facilitate the medication management of depression and other psychiatric disorders when possible by collaborating with the prescribing HCV physicians.
  Arms: Integrated Care

SUMMARY:
To determine the effect of an integrated care protocol on antiviral treatment and sustained virologic response (SVR) rates following initiation of direct acting antiviral therapies (DAA) treatments in 2011.

DETAILED DESCRIPTION:
Background and aims: Approval of direct acting antiviral (DAA) therapies in 2011 initiated a new era of more effective treatments for hepatitis C (HCV). The impact of more effective therapies on patient access to treatment is unknown. Integrated Care (IC) involving patient case management may overcome barriers to treatment access imposed by psychiatric and substance use disorders (SUD).

Methods: Prospective, randomized trial at a single medical center. Patients with HCV at risk for active psychiatric and SUD between Jan 2012 and Jan 2013 were recruited and randomized to IC or Usual Care (UC). A mid-level mental health practitioner was placed in the IC clinic and provided brief mental health care and case management.

ELIGIBILITY:
Inclusion Criteria:

* Patients with HCV infection who were referred to the VA HCV clinic and who received the usual initial evaluation in the clinic
* All patients 18 and 75 years old with confirmed HCV infection
* Patients were required to be classified as "high risk candidates for antiviral treatment" on any one of a set of screening measure in order to participate
* Screening measures and cutoffs for inclusion were depression:

  * Beck Depression Inventory: (BDI) > 10
  * Alcohol use: Alcohol Use Disorders Identification Test (AUDIT-C) > 4
  * PTSD: VA Primary Care PTSD Screen = endorsement of three or more items or any single endorsement of item #3
  * Drug use: Drug Use Questionnaire = self-reported drug/alcohol use within 6 months prior to screen

Exclusion Criteria:

* Lacked a confirmed test of HCV RNA
* Had HIV/HCV co-infection and received care at San Diego or Palo Alto sites (these patients were treated in a separate clinic)
* Had Hepatitis B (HBV) co-infection
* Had decompensated liver disease with active or recent encephalopathy, variceal bleeding, or ascites or Child-Pugh class B or C
* Had other significant near term life-threatening diseases
* Were treatment non-responders with pegylated Interferon plus ribavirin

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 83 (Actual)
Dates: Start 2012-01; Primary Completion 2013-01 (Actual); Study Completion 2014-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Samuel B Ho, MD, Principal Investigator — VA San Diego Healthcare System, San Diego, CA
Locations (1):
- VA San Diego Healthcare System, San Diego, CA, San Diego, California, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 83 patients were consented but only 79 were randomized. 4 participants were withdrawn.
Period: Overall Study
Arm/Group | Integrated Care | Usual Care
Started | 40 | 39
Completed | 40 | 39
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Integrated Care | Usual Care | Total
Number analyzed (Participants) | 40 | 39 | 79
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.0 (8.7) | 57.4 (7.7) | 55.7 (8.4)
Gender [Number; unit: participants] — Gender data was not collected from 4 participants.
  participants
    Female | 0 | 0 | 0
    Male | 37 | 38 | 75
Race/Ethnicity, Customized [Number; unit: participants]
  African American or Black | 7 | 12 | 19
  Native American | 0 | 1 | 1
  Hispanic | 7 | 4 | 11
  Asian/Pacific Islander | 1 | 0 | 1
  White | 25 | 22 | 47
Region of Enrollment [Number; unit: participants]
  United States | 40 | 39 | 79
Marital Status [Number; unit: participants]
  Single | 11 | 9 | 20
  Married or widowed | 11 | 14 | 25
  Separated or Divorced | 18 | 15 | 33
  Missing | 0 | 1 | 1
Education [Number; unit: participants]
  Grade 1 to 8 | 0 | 1 | 1
  Grade 9 to 11 | 2 | 2 | 4
  High school/GED | 12 | 6 | 18
  Some College | 21 | 22 | 43
  College Grad | 2 | 4 | 6
  Post Grad | 0 | 1 | 1
  Missing | 3 | 3 | 6
Employment [Number; unit: participants]
  Full and Part time | 4 | 5 | 9
  Unemployed | 13 | 15 | 28
  Disabled | 15 | 14 | 29
  Retired or Volunteer | 7 | 4 | 11
  Missing | 1 | 1 | 2
Homeless in last 5 years [Number; unit: participants]
  Homeless in the last 5 years | 18 | 20 | 38
  Missing | 3 | 5 | 8
  Not Homeless | 19 | 14 | 33
BMI [Mean (Standard Deviation); unit: Kilograms/m2] | 29.0 (5.8) | 28.6 (5.3) | 28.8 (5.5)

OUTCOME MEASURES:

1. Primary Outcome: Sustained Viral Response (SVR)
Description: The primary outcome for the study was the proportion of patients that achieve an SVR. Patient adherence to completing the prescribed therapy and SVR were both tracked with medical records. Viral load at 4, 12-and 24-weeks during treatment initiation have been shown to predict final SVR. Final SVR data consists of viral tests conducted at 6 months after the termination of therapy.
Time Frame: up to 24 weeks
Measure: Number; unit: percentage of Participants
Arm/Group | Integrated Care | Usual Care
Number analyzed (Participants) | 40 | 39
percentage of Participants | 30 | 12.8
Statistical Analysis 1: Comparison: Integrated Care vs Usual Care; Test type: Superiority or Other; p = 0.07, Regression, Linear; Multivariable Regression Analysis; Odds Ratio (OR) = 2.91, 95% CI 2-sided [0.92 to 9.27]

2. Secondary Outcome: Percentage of Participants With Treatment Initiation and Completion
Description: The main secondary outcomes for the study include rates of Interferon-based treatment initiation and completion. Treatment data from the HCV clinics were reviewed for each patient at each site. Participants who a) filled at least one prescription for Interferon and ribavirin, and b) had at least one treatment-related physician visit with a medical record note stating they began taking the medications were deemed to have initiated antiviral treatment. Patients were considered to have completed treatment if they a) were prescribed and received the full course of antiviral treatment recommended by their HCV physician, and b) had at least one medical record note stating they had completed treatment.
Time Frame: up to 24 weeks
Measure: Number; unit: percentage of Particpants
Arm/Group | Integrated Care | Usual Care
Number analyzed (Participants) | 40 | 39
percentage of Particpants | 45 | 23.1

3. Secondary Outcome: Percentage of Participants That Completed Planned Duration of Treatment Using a Cutoff of 80%
Description: Patients were considered to have completed treatment if they a) were prescribed and received the full course of antiviral treatment recommended by their HCV physician, and b) had at least one medical record note stating they had completed treatment.
Time Frame: up to 24 weeks
Measure: Number; unit: percentage of participants
Arm/Group | Integrated Care | Usual Care
Number analyzed (Participants) | 40 | 39
percentage of participants | 78 | 63

ADVERSE EVENTS:
Arm/Group | Integrated Care | Usual Care
Serious Adverse Events (participants affected / at risk) | 8/40 | 6/39
Other Adverse Events (participants affected / at risk) | 0/40 | 0/39
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Integrated Care (N=40) | Usual Care (N=39)
Hospitalization (General disorders) | 8 | 6 — Unknown Cause
Death (General disorders) | 1 | 3 — Unknown cause
Death (Cardiac disorders) | 0 | 1 — Heart attack caused by long term substance abuse
Death (Respiratory, thoracic and mediastinal disorders) | 0 | 1 — Pulseless electrical activity most likely secondary to pulmonary emboli.
Death (General disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes